CLINICAL TRIAL: NCT03534843
Title: A Comparison Between Child-Pugh and Albumin-Bilirubin Scores in Patients With Spontaneous Rupture of Hepatocellular Carcinoma: A Retrospective Study
Brief Title: A Comparison Between Child-Pugh and Albumin-Bilirubin Scores
Status: Completed | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaoping Chen, Professor, Huazhong University of Science and Technology
Other Study IDs: Chenxp011
Record Dates: First submitted 2018-05-12; First posted 2018-05-23 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Rupture, Spontaneous; Rupture Liver; Hepatocellular Carcinoma; Hepatic Impairment
Keywords: Spontaneous rupture; survival; hepatocellular carcinoma; Child-Pugh; Albumin-bilirubin
MeSH Terms: conditions — Rupture, Spontaneous; Carcinoma, Hepatocellular | interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgical treatment: Patients who received liver resection or palliative surgery, such as microwave coagulation therapy, hepatic artery ligation, or suturing ligation.
  Interventions: Procedure: Liver resection
- Non-surgical treatment: Patients who received transcatheter arterial embolization (or transcatheter arterial chemoembolization) or conservative treatment
  Interventions: Other: Transcatheter arterial embolization

INTERVENTIONS:
Procedure: Liver resection — Liver resection was comprised of single or multiple liver resections aiming to excise all macroscopic tumors.
  Groups: Surgical treatment
Other: Transcatheter arterial embolization — Transcatheter arterial embolization or transcatheter arterial chemoembolization can localize the bleeding point and provide interventional embolization.
  Groups: Non-surgical treatment

SUMMARY:
To compare Child-Pugh and Albumin-Bilirubin scores in patients with spontaneous rupture of hepatocellular carcinoma

DETAILED DESCRIPTION:
To compare Child-Pugh and Albumin-Bilirubin scores in patients with spontaneous rupture of hepatocellular carcinoma. And to determine which is better in predicting long-term survival and short-term survival.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed as hepatocellular carcinoma pathologically; had a tumor rupture confirmed by Intraperitoneal exploration or clinical signs and symptoms in combination with imaging examination.

Exclusion Criteria:

* Be diagnosed as not hepatocellular carcinoma pathologically；had repeated transcatheter arterial chemoembolization(TACE) or a long history (more than 1 year) of cancer treatment; loss of follow up or without complete data.

Ages: 15 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From January 2005 to August 2015, all patients complied with the criteria mentioned above who received surgical treatment or non-surgical treatment at the investigator's center were included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2015-08-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Overall survival of all patients | 5 years
  Overall survival of all patients among different Child-Pugh and albumin-bilirubin scores

SECONDARY OUTCOMES:
Short-term mortality of all patients | Ninety days
  Ninety-day mortality of all patients among different Child-Pugh and albumin-bilirubin scores
Short-term mortality of surgical subgroup | Ninety days
  Ninety-day mortality of the surgical subgroup among different Child-Pugh and albumin-bilirubin scores
Short-term mortality of non-surgical subgroup | Ninety days
  Ninety-day mortality of the non-surgical subgroup among different Child-Pugh and albumin-bilirubin scores

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-ping Chen, Prof. PHD, Study Chair — Huazhong University of Science and Technology

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wu JJ, Zhang ZG, Zhu P, Mba'nbo-Koumpa AA, Zhang BX, Chen XP, Shu C, Zhang WG, Feng RJ, Li GX. Comparative liver function models for ruptured hepatocellular carcinoma: A 10-year single center experience. Asian J Surg. 2019 Sep;42(9):874-882. doi: 10.1016/j.asjsur.2018.12.015. Epub 2019 Jan 28. PMID 30704966